CLINICAL TRIAL: NCT06191315
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Efficacy and Longterm Safety of Dupilumab in Children 2 to <6 Years of Age With Uncontrolled Asthma and/or Recurrent Severe Asthmatic Wheeze
Brief Title: Efficacy and Safety of Subcutaneous Dupilumab in Participants With Asthma/Asthmatic Wheeze Aged 2 to <6 Years (LIBERTY ASTHMA TREKIDS)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC14771; 2023-504331-41 (Registry Identifier: CTIS); U1111-1246-7432 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Wheezing; Asthma
MeSH Terms: conditions — Respiratory Sounds; Asthma | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dupilumab (double-blind period) (Experimental): Dupilumab subcutaneous injection as per protocol
  Interventions: Drug: Dupilumab
- Placebo (Placebo Comparator): Placebo matching dupilumab subcutaneous injection as per protocol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab — Pharmaceutical form: Injection solution Route of administration: Subcutaneous
  Other Names: SAR231893; Dupixent
  Arms: Dupilumab (double-blind period)
Drug: Placebo — Pharmaceutical form: Injection solution Route of administration: Subcutaneous
  Arms: Placebo

SUMMARY:
This is a parallel, Phase 3, 2-arm study to evaluate the efficacy and long-term safety of dupilumab treatment in children 2 to <6 years of age with uncontrolled asthma and/or recurrent severe asthmatic wheeze. The study will be conducted in 2 parts. Part A will be a 52-week, randomized, double-blind, placebo-controlled study to assess the safety and efficacy of dupilumab in children aged 2 to <6 years old with uncontrolled asthma and/or recurrent severe asthmatic wheeze. At the end of Part A, all eligible participants will be offered participation in Part B, an optional open-label extension phase.

Study details include:

Part A:

The study duration of part A will be up to 68 weeks consisting of a 4-week Screening, a 52week treatment period, and a 12-week post-treatment follow-up period. For participants who will chose to participate in Part B, the study duration will be up to 120 weeks (additional 52-week treatment period).

Part B:

For participants who will choose to participate in Part B, the study duration will be up to 120 weeks (Part A [4-week Screening and a 52-week treatment period] plus additional 52-week treatment period and a 12-week post-treatment follow-up period).

DETAILED DESCRIPTION:
The duration per participant is up to 120 Weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 2 to <6 years of age
* Diagnosis of asthma or recurrent severe asthmatic wheeze that is not controlled with chronic ICS for at least 3 months with stable use of at least low dose ICS for ≥1 month prior to Screening Visit 1 with evidence of uncontrolled asthma and/or recurrent severe asthmatic wheeze.
* At least one additional major criterion from the modified asthma predictive index:

  1. Physician diagnosed Atopic Dermatitis,
  2. Allergic sensitization to at least 1 aeroallergen (with a positive serum IgE defined as a value ≥0.35 kU/L).

     OR 2 minor criteria:
  3. Wheezing unrelated to colds,
  4. Peripheral blood eosinophilia ≥4%,
  5. Allergic sensitization to milk, eggs, or peanuts (defined by serum specific IgE >0.35 kU/L.
* Parent(s)/caregiver(s)/legal guardian(s) willing and able to comply with clinic visits and study-related procedures.
* Parent(s)/caregiver(s)/legal guardian(s) able to understand the study requirements.
* Participants/parent(s)/caregiver(s)/legal guardian(s), as appropriate, must be able to understand and complete study-related questionnaires
* Body weight at screening and randomization >5 kg and <30 kg.
* Parents or caregivers or legal guardian capable of giving signed informed consent.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Severe asthma with the need for chronic oral/systemic corticosteroid use (>1 month continuous) at the time of screening enrollment.
* History of a systemic hypersensitivity reaction or anaphylaxis to biologic therapy, including any excipient.
* History of prematurity (<34 weeks gestation).
* Any other chronic lung disease that would impair lung function (eg, cystic fibrosis, bronchopulmonary dysplasia) or chronic lung disease of prematurity or need for oxygen for more than 5 days in the neonatal period.
* History of life-threatening asthma (eg, requiring intubation).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2028-12-21 (Estimated); Study Completion 2028-12-21 (Estimated)

PRIMARY OUTCOMES:
Part A: Annualized rate of severe asthma exacerbations during the 52-week treatment period | Baseline through Week 52
  Annualized rate of severe asthma exacerbations during the 52-week treatment period.
Part B: Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events of special interest (AESIs), and AEs leading to permanent treatment discontinuation | Week 52 through Week 116
  Incidence of TEAEs, SAEs, AESIs, and AEs leading to permanent treatment discontinuation.

SECONDARY OUTCOMES:
Part A: Annualized rate of hospitalization, ER or urgent care visit for asthma exacerbation during the 52week treatment period. | Baseline through Week 52
Part A: Annualized rate of moderate asthma exacerbations during the 52-week treatment period | Baseline through Week 52
  Annualized rate of moderate asthma exacerbations during the 52-week treatment period.
Part A: Cumulative ICS dose during the 52-week treatment period | Baseline through Week 52
Part A: Change from baseline in weekly average use of reliever medication during the 52-week treatment period | Baseline to Week 52
Part A: Mean number of days without asthma symptoms (DWAS) using the Pediatric Asthma Caregiver Diary (PACD) during the 52-week treatment period | Baseline through Week 52
  A day without asthma symptoms (DWAS) is defined as a day without any asthma symptoms, β-agonist use, oral steroid use, or need for urgent asthma care. The PACD consists of a daytime and overnight record. The daytime asthma symptom questions are scored on a 6-point scale from 0 (no symptoms/interference) to 5 (very severe symptoms/interference). The overnight questions are scored on a 5-point scale from 0 (no overnight cough and caregiver not disturbed at all) to 4 (coughed all night and disturbed all night).
Part A: Change from baseline to Week 52 in daytime symptom score using the daytime record of PACD | Baseline to Week 52
  The PACD consists of a daytime and overnight record. The daytime asthma symptom questions are scored on a 6-point scale from 0 (no symptoms/interference) to 5 (very severe symptoms/interference).
Part A: Incidence of TEAEs, SAEs, AESIs, and AEs leading to permanent treatment discontinuation | Baseline through Week 52
Part A: Change from baseline to Week 52 in Pediatric Quality of Life Inventory (PedsQL) 4.0 Generic Scale | Baseline to Week 52
  PedsQL measures health-related quality of life (HRQOL) in healthy children and adolescents and those with acute and chronic health conditions. Scores range 0-100 with higher scores indicate better HRQOL.
Part A: Caregiver Global Impression of Change in their child's asthma control (CGI-change in asthma control) at Week 52 | Week 52
  CGI-change in asthma control is a 1-item questionnaire that asks the caregiver to provide the overall assessment of change of their child's asthma control on a 7-point scale, compared to just before he/she started taking the study treatment. Response choices are: 0 = "Very much better", 1 ="Moderately better", 2 = "A little better", 3 = "No change", 4 = "A little worse", 5 = "Moderately worse", 6 = "Very much worse".
Part A: Physician Global Assessment of Change of the child's asthma control (PGA-change in asthma control) at Week 52 | Week 52
  The Physician Global Assessment of Change of Asthma (PGA-change in asthma control) is a 1 item questionnaire that asks the physician to provide the overall assessment of change in the child's asthma control on a 7-point scale, compared to just before he/she started taking the study treatment. Response choices are: 0 = "Very much better", 1 = "Moderately better", 2 ="A little better", 3 = "No change", 4 = "A little worse", 5 = "Moderately worse", 6 = "Very much worse".
Part A: Change from baseline to Week 52 in Caregiver Global Impression of their child's asthma control (CGI-asthma control) | Baseline to Week 52
  The Caregiver Global Impression of asthma control (CGI-Asthma Control) is a 1-item questionnaire that asks caregiver to provide the assessment of their child's asthma control over the past 7 days, on a 4-point scale for the past week. Response choices are: 1 = "Not controlled", 2 = "Somewhat controlled", 3 = "Moderately controlled", 4 = "Well controlled".
Part A: Change from baseline to Week 52 in Caregiver Global Impression of their child's asthma severity (CGI-asthma severity) | Baseline to Week 52
  The Caregiver Global Impression of asthma severity (CGI-Asthma Severity) is a 1-item questionnaire that asks caregivers to provide the assessment of their child's asthma control over the past 7 days, on a 4-point scale for the past week. Response choices are: 1 = "None", 2 = "Mild", 3 = "Moderate", 4 = "Severe".
Part A: Change from baseline to Week 52 in Physician Global Assessment of the child's asthma control (PGA-asthma control). | Baseline to Week 52
  The Physician Global Assessment of asthma control is a 1-item questionnaire that asks physicians to assess the control of the child's asthma in the past 7 days on a 4 point scale for the past week. Response choices are: 1 = "Not controlled", 2 = "Somewhat controlled", 3 = "Moderately controlled", 4 = "Well controlled".
Part A: Change from baseline to Week 52 in Test for Respiratory and Asthma Control in Kids (TRACK) | Baseline to Week 52
  TRACK is a validated questionnaire for caregiver completion for preschool aged children with symptoms consistent with asthma. The total score range of 0 to 100. Higher scores indicated better asthma control.
Part A: Change from baseline in blood eosinophil level at Weeks 24 and 52 | Baseline to Week 24 and 52
Part A: Concentration of dupilumab in serum over time during the 52-week treatment period | Baseline through Week 52
Part A: Incidence of treatment-emergent anti-drug antibody (ADA) against dupilumab over time | Baseline through Week 52
Part A: IgG response to any vaccination for tetanus, diphtheria and pertussis and antibody for influenza (HAI antibody titers) vaccine administered according to vaccination schedule during the 52-week treatment period | Baseline through Week 52
Part B: Annualized rate of severe asthma exacerbations events during the 52-week Part B treatment period | Week 52 through Week 104
  Annualized rate of severe asthma exacerbations events during the 52-week Part B treatment period.
Part B Concentration of dupilumab in serum over time during the 52-week Part B treatment period | Week 52 through Week 104
Part B: Incidence of treatment-emergent anti-drug antibodies (ADAs) against dupilumab over time | Week 52 through Week 104

CONTACTS AND LOCATIONS:
Locations (75):
- United States (14):
  - Phoenix Children's Hospital- Site Number : 8400001, Phoenix, Arizona
  - Allervie Clinical Research - Destin- Site Number : 8400016, Destin, Florida
  - EMDA Clinical Research- Site Number : 8400026, Miami, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago- Site Number : 8400011, Chicago, Illinois
  - Allergy and Asthma Specialist- Site Number : 8400002, Owensboro, Kentucky
  - Mayo Clinic in Rochester - Minnesota- Site Number : 8400008, Rochester, Minnesota
  - UBMD Pediatrics- Site Number : 8400013, Buffalo, New York
  - Boston Children's Health Physicians - Hawthorne- Site Number : 8400010, Hawthorne, New York
  - UNC Children's Hospital- Site Number : 8400005, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center- Site Number : 8400004, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center- Site Number : 8400015, Cleveland, Ohio
  - Vanderbilt University Medical Center- Site Number : 8400024, Nashville, Tennessee
  - South Texas Medical Research Institute - TTS Research- Site Number : 8400022, Boerne, Texas
  - Texas Children's Hospital - Baylor - PIN- Site Number : 8400027, Houston, Texas
- Argentina (8):
  - Investigational Site Number : 0320005, Rosario, Santa Fe Province
  - Investigational Site Number : 0320008, Buenos Aires
  - Investigational Site Number : 0320003, Buenos Aires
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320009, Corrientes
  - Investigational Site Number : 0320006, Córdoba
  - Investigational Site Number : 0320004, Mendoza
- Brazil (4):
  - Instituto de Medicina Integral Professor Fernando Figueira- Site Number : 0760006, Recife, Pernambuco
  - Hospital Ernesto Dornelles- Site Number : 0760004, Porto Alegre, Rio Grande do Sul
  - Clinica de Alergia Martti Antila- Site Number : 0760002, Sorocaba, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo- Site Number : 0760001, São Paulo
- Canada (6):
  - Investigational Site Number : 1240002, Edmonton, Alberta
  - Investigational Site Number : 1240001, Vancouver, British Columbia
  - Investigational Site Number : 1240008, Burlington, Ontario
  - Investigational Site Number : 1240007, Hamilton, Ontario
  - Investigational Site Number : 1240006, Montreal, Quebec
  - Investigational Site Number : 1240005, Sherbrooke, Quebec
- Investigational Site Number : 2030001, Prague, Czechia
- France (5):
  - Investigational Site Number : 2500005, Créteil
  - Investigational Site Number : 2500001, Lille
  - Investigational Site Number : 2500004, Nice
  - Investigational Site Number : 2500002, Paris
  - Investigational Site Number : 2500003, Paris
- Germany (3):
  - Investigational Site Number : 2760002, Düsseldorf
  - Investigational Site Number : 2760004, Frankfurt
  - Investigational Site Number : 2760001, Leipzig
- Greece (2):
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000003, Athens
- Hungary (4):
  - Investigational Site Number : 3480005, Budapest
  - Investigational Site Number : 3480004, Debrecen
  - Investigational Site Number : 3480002, Székesfehérvár
  - Investigational Site Number : 3480001, Szigetvár
- Italy (5):
  - Buzzi Children's Hospital - Investigational Site Number : 3800003, Milan, Lombardy
  - Investigational Site Number : 3800005, Padua, Padova
  - Ospedale Pediatrico Bambino Gesù - Investigational Site Number : 3800002, Rome, Roma
  - AOU Luigi Vanvitelli - Investigational Site Number : 3800004, Napoli
  - Fondazione IRCCS Policlinico San Matteo - Investigational Site Number : 3800001, Pavia
- Japan (5):
  - Investigational Site Number : 3920006, Isehara, Kanagawa
  - Investigational Site Number : 3920004, Tsu, Mie-ken
  - Investigational Site Number : 3920003, Ureshino, Saga-ken
  - Investigational Site Number : 3920002, Fukuoka
  - Investigational Site Number : 3920001, Fukuoka
- Mexico (3):
  - Investigational Site Number : 4840001, San Juan del Río, Querétaro
  - Investigational Site Number : 4840004, Durango
  - Investigational Site Number : 4840002, Veracruz
- Investigational Site Number : 5280001, Rotterdam, Netherlands
- Poland (3):
  - Investigational Site Number : 6160004, Tarnów, Lesser Poland Voivodeship
  - Investigational Site Number : 6160001, Lodz, Lódzkie
  - Investigational Site Number : 6160003, Warsaw, Masovian Voivodeship
- Spain (7):
  - Investigational Site Number : 7240003, Santiago de Compostela, A Coruña [La Coruña]
  - Investigational Site Number : 7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240007, Esplugues de Llobregat, Barcelona [Barcelona]
  - Investigational Site Number : 7240002, Sabadell, Barcelona [Barcelona]
  - Investigational Site Number : 7240006, Jerez de la Frontera, Cádiz
  - Investigational Site Number : 7240005, Madrid
  - Investigational Site Number : 7240004, Valencia
- United Kingdom (4):
  - Investigational Site Number : 8260003, Birmingham, England
  - Investigational Site Number : 8260002, Leicester, Leicestershire
  - Investigational Site Number : 8260001, London, London, City of
  - Investigational Site Number : 8260004, Bradford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC14771 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25594&tenant=MT_SNY_9011